CLINICAL TRIAL: NCT05916716
Title: Use of a Novel Volume-stable Collagen Matrix (VCMX) in the Treatment of Single Gingival Recession Associated With Non-carious Cervical Lesion Partially Restored. A Randomized Clinical Trial
Brief Title: Use of a Novel Volume-stable Collagen Matrix (VCMX) in the Treatment of Single Gingival Recession Associated With Non-carious Cervical Lesion Partially Restored
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Associate Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UEPJMF 13
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Gingival Recession, Localized; Tooth Abrasion
Keywords: Gingival Recession; Tooth Abrasion; Biomaterials
MeSH Terms: conditions — Gingival Recession; Tooth Abrasion | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR+CAF (Active Comparator): Partial restoration will be performed, and its apical margin will be placed 1 mm beyond the estimated position of the cementoenamel junction. Patients enrolled in this group will receive a coronally advanced flap (CAF). Two horizontal incisions will be performed at the papilla base united by an intrasulcular incision around the tooth. In sequence, releasing incisions will be designed and a split-full-split flap will be raised beyond the mucogingival junction. Sling sutures will be placed to stabilize the flap margin 2 mm coronal to CEJ, followed by interrupted sutures to close the releasing incisions.
  Interventions: Procedure: Restorative procedure; Procedure: Coronally Advanced Flap (CAF).; Drug: Sodium dipyrone
- PR + CAF + VCMX (Experimental): Partial restoration will be performed, and its apical margin will be placed 1 mm beyond the estimated position of the cementoenamel junction. Patients enrolled in this group will receive a coronally advanced flap (CAF) associated with a volume-stable collagen matrix (VCMX). Two horizontal incisions will be performed at the papilla base united by an intrasulcular incision around the tooth. In sequence, releasing incisions will be designed and a split-full-split flap will be raised beyond the mucogingival junction. In sequence, VCMX will be cut according to the recession defect and moistened with saline solution. The biomaterial will be placed at the cementoenamel junction level and stabilized in the adjacent surgery papillae by interrupted sutures. Then, sling sutures will be placed to stabilize the flap margin 2 mm coronal to CEJ, followed by interrupted sutures to close the releasing incisions.
  Interventions: Procedure: Restorative procedure; Procedure: Coronally Advanced Flap (CAF).; Device: Volume-stable collagen matrix (VCMX); Drug: Amoxicillin 500mg; Drug: Sodium dipyrone

INTERVENTIONS:
Procedure: Restorative procedure — Under local anesthesia, a rubber dam isolation will be placed at the site and a coronal bevel will be performed at the incisal margin of the NCCL allowing a correct tooth emergence profile. In sequence, acid etching with 35% phosphoric acid will be applied to the area and washed for 30 seconds with a water-air jet. The lesion will be dried with sterile cotton pellets to prevent dehydration. Active application of the adhesive will be performed for 20 seconds, followed by light curing for 30 seconds. The apical margin of the restoration will be placed 1 mm beyond the estimated position of the cementoenamel junction(CEJ) in order to rebuild only the anatomical part of the crown destroyed by the NCCL and 1 mm of the root surface to give the appropriate emergence profile. After rubber dam removal, the restoration will be finished with ultrafine-grained burs, and 48 hours after the restoration procedure, polishing will be completed with diamond paste and felt discs.
Procedure: Coronally Advanced Flap (CAF). — Two horizontal incisions will be performed at the papilla base united by an intrasulcular incision around the tooth. In sequence, releasing incisions will be designed and a split-full-split flap will be raised beyond the mucogingival junction. Then, sling sutures will be placed to stabilize the flap margin 2 mm coronal to CEJ, followed by interrupted sutures to close the releasing incisions.
Device: Volume-stable collagen matrix (VCMX) — VCMX will be cut according to the recession defect and moistened with saline solution. The biomaterial will be placed at the cementoenamel junction (CEJ) level and stabilized in the adjacent surgical papillae by interrupted sutures.
  Arms: PR + CAF + VCMX
Drug: Amoxicillin 500mg — Participants enrolled in the PR +CAF+VCMX will be instructed to take amoxicillin 500mg (8 hours/8 hours, during 7 days) after the surgical procedures.
  Other Names: Post operative care
  Arms: PR + CAF + VCMX
Drug: Sodium dipyrone — All participants will be instructed to take 500 mg sodium dipyrone just in case of pain.
  Other Names: Post operative care

SUMMARY:
Gingival recessions (GR) are often associated with non-carious cervical lesions (NCCL), resulting, thus, in a combined defect. This mucogingival condition has a different treatment prognosis when compared with a GR without wearing surface associated and frequently requires a surgical-restorative approach to achieve better esthetics and functional results. A limited number of clinical studies assessed different multidisciplinary protocols for the management of single combined defects and there is evidence that the use of dental materials does not harm the periodontal tissues and does not influence the root coverage obtained by means of subepithelial connective tissue graft (CTG). Although the association between coronally advanced flap (CAF) and CTG provides more predictable and stable outcomes in the long term, its use is related to some drawbacks. Different biomaterials have been developed to overcome these limitations as a possible alternative to autogenous graft. However, despite its potential, there is a lack of studies evaluating its use in treating this type of condition. Thus, this study aims to assess from a clinical and esthetics point of view and patient-centered outcomes, the use of a new collagen matrix (Geistlich Fibro-Gide®) associated with CAF for the management of single combined defects. For such purpose, 50 patients with single RT1 gingival recessions associated with NCCL will be enrolled and randomly allocated to one of the following groups: control group (n=25), partial restoration of cervical lesion and coronally advanced flap for root coverage (PR+CAF) and test group (n=25), partial restoration of cervical lesion and coronally advanced flap associated with volume stable collagen matrix (PR+CAF+VCMX). The two groups will be compared regarding the clinical parameters, among which bleeding on probing (BOP), biofilm accumulation (IP), clinical attachment level (CAL), recession reduction (RecRed), and the percentage of combined defect coverage (%CDC). Patient-reported outcomes such as post-surgery pain and discomfort, time to recover, the decrease of dentin hypersensitive, and aesthetics will be gathered. A professional assessment will be carried out regarding the aesthetic parameters. All these evaluations will be performed at the baseline and three and six months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* adult > 20 years old;
* systemically healthy
* no signs of active periodontal disease;
* full-mouth plaque and bleeding score ≤20%;
* Gingival recession type RT1 associated with NCCL B+ on a vital canine or premolar;

Exclusion Criteria:

* Patients who had had periodontal surgery on the study area;
* Smokers patients;
* Pregnant or lactating patients;
* Ongoing orthodontic treatment;
* Patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Recession reduction (RecRed) | 180 days
  Difference between the final depth of gingival recession in millimeters and gingival margin initial position in millimeters measured through a periodontal probe.

SECONDARY OUTCOMES:
Dentine hypersensitivity | 180 days
  Root sensitivity assessemnt with the air blow test and measurement with a visual analog scale (VAS).
Patient-centered esthetic evaluation | 180 days
  Using a visual analog scale (VAS), patients will be able to report their opinion regarding esthetic
Oral Health Impact Profile | 14 days
  Will be evaluated from a questionnaire with 14 questions based on 7 domains: functional limitations, physical pain, psychological discomfort, physical disability, psychological deficiency and social deficiency. The patient should respond to the questions within 14 days after the surgical procedure, performing a postoperative diary. For each question an answer must be given, represented in numbers, being: 0- Never; 1- Almost never; 2-Occasionally; 3-Quite frequent; 4-Very common; 5-I do not know (Tonetti MS et al. 2017)
Patient Discomfort | 14 days
  By a visual analogic scale (VAS) of 100 mm to assess discomfort, patients will report pain diary during the 14 days after surgery. Scale extremes will be "no pain" to "extreme." (Tonetti et al. 2017).
Number of analgesics | 14 days
  Number of analgesics used during 14 days after the procedure will be reported at the same postoperative diary (Tonetti et al. 2017).
Percentage of Complete Combined Defect Coverage (%CDC) | 180 days
  This assement is calculated as follow: (RecRed x 100)/CD
Modification of the Root Coverage Esthetic Score (MRES) | 180 days
  Professional aesthetic score which evaluates six variables. The variables are :(1) the marginal tissue contour (MTC); (2) Soft tissue texture (STT); (3) mucogingival junction alignment (MGJ); (4) Gingival color (GC) and (5) Restoration/cervical lesion color (R/CLC).
Clinical Parameters | 180 days
  Probing Depth (PD); Relative Gingival Recession (RGR); Relative Clinical Attachment level (RCAL); Keratinized tissue width (KTW); Keratinized tissue thickness (KTT).

CONTACTS AND LOCATIONS:
Locations (1):
- Sao Paulo State University, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Santamaria MP, Miguel MMV, Rossato A, Bonafe ACF, Ferraz LFF, Dos Santos LM, Mathias-Santamaria IF. New Volume-Stable Collagen Matrix and Modified Coronally Advanced Flap to Treat Multiple Gingival Recessions Associated With Partially Restored Non-Carious Cervical Lesions: A Case Report. Clin Adv Periodontics. 2022 Jun;12(2):69-74. doi: 10.1002/cap.10142. Epub 2020 Dec 16. PMID 33289326
- [Background] Santamaria MP, Mathias-Santamaria IF, Ferraz LFF, Casarin RCV, Romito GA, Sallum EA, Pini-Prato GP, Casati MZ. Rethinking the decision-making process to treat gingival recession associated with non-carious cervical lesions. Braz Oral Res. 2021 Sep 24;35(Supp 2):e096. doi: 10.1590/1807-3107bor-2021.vol35.0096. eCollection 2021. PMID 34586210
- [Background] Santamaria MP, Fernandes-Dias SB, Araujo CF, Lucas da Silva Neves F, Mathias IF, Rebelato Bechara Andere NM, Neves Jardini MA. 2-Year Assessment of Tissue Biostimulation With Low-Level Laser on the Outcomes of Connective Tissue Graft in the Treatment of Single Gingival Recession: A Randomized Clinical Trial. J Periodontol. 2017 Apr;88(4):320-328. doi: 10.1902/jop.2016.160391. Epub 2016 Nov 11. PMID 27834120
- [Background] de Sanctis M, Zucchelli G. Coronally advanced flap: a modified surgical approach for isolated recession-type defects: three-year results. J Clin Periodontol. 2007 Mar;34(3):262-8. doi: 10.1111/j.1600-051X.2006.01039.x. PMID 17309597
- [Result] Mathias-Santamaria IF, Silveira CA, Rossato A, Sampaio de Melo MA, Bresciani E, Santamaria MP. Single gingival recession associated with non-carious cervical lesion treated by partial restoration and coronally advanced flap with or without xenogenous collagen matrix: A randomized clinical trial evaluating the coverage procedures and restorative protocol. J Periodontol. 2022 Apr;93(4):504-514. doi: 10.1002/JPER.21-0358. Epub 2021 Aug 21. PMID 34310715
- [Result] Stefanini M, Mounssif I, Barootchi S, Tavelli L, Wang HL, Zucchelli G. An exploratory clinical study evaluating safety and performance of a volume-stable collagen matrix with coronally advanced flap for single gingival recession treatment. Clin Oral Investig. 2020 Sep;24(9):3181-3191. doi: 10.1007/s00784-019-03192-5. Epub 2020 May 2. PMID 32361892
- [Derived] Santamaria MP, Miguel MMV, Rossato A, Bonafe ACF, de Souza IV, Martins TM, Nunes MP, Mathias-Santamaria IF. Volume-stable collagen matrix to treat gingival recession associated with non-carious cervical lesions: Randomized clinical trial. J Periodontol. 2025 Aug 21. doi: 10.1002/jper.11386. Online ahead of print. PMID 40838330